CLINICAL TRIAL: NCT02247557
Title: Intravesical Instillation of Liposome Encapsulated Botulinum Toxin A (Lipotoxin) in Treatment of Interstitial Cystitis - a Randomized, Double-blind, Placebo-controlled, Prospective Study
Brief Title: Intravesical Instillation of Liposome Encapsulated Botulinum Toxin A (Lipotoxin) in Treatment of Interstitial Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Director of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCGHUROL011
Record Dates: First submitted 2014-09-15; First posted 2014-09-25 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Interstitial Cystitis
Keywords: IC/PBS; VAS; Botulinum Toxin A; Lipotoxin
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Liposomes; Botulinum Toxins, Type A; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled physician initiated study enrolled patients with refractory IC/BPS. Patients were assigned to intravesical instillation of lipotoxin (onabotulinumtoxinA 200 U with 80mg sphingomyelin), onabotulinumtoxinA 200 U in normal saline, or normal saline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants, investigators and care providers do not know which regimen is given to patients of the three arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Liposome encapsulated BoNT-A (Experimental): Liposome encapsulated BoNT-A ( mixed BOTOX 200U/10ml in Liposome 80mg/40ml) in single intravesical instillation
  Interventions: Drug: Liposome encapsulated BoNT-A
- Group B: BoNT-A 200 U in Normal saline (Experimental): BOTOX 200U in normal saline (BoNT-A/NS) 50ml in single intravesical instillation
  Interventions: Drug: BOTOX 200U in normal saline
- Group C: Normal saline (Placebo Comparator): Normal saline (N/S) 50ml in single intravesical instillation
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Liposome encapsulated BoNT-A — Liposome encapsulated BoNT-A ( mixed BOTOX 200U/10ml in Liposome 80mg/40ml) in single intravesical instillation
  Other Names: Liposome; onabotulinumtoxinA 200U
  Arms: Group A: Liposome encapsulated BoNT-A
Drug: BOTOX 200U in normal saline — BOTOX 200U in normal saline (BoNT-A/NS) 50ml in single intravesical instillation
  Other Names: onabotulinumtoxinA 200U
  Arms: Group B: BoNT-A 200 U in Normal saline
Drug: Normal saline — Normal saline (N/S) 50ml in single intravesical instillation
  Other Names: Saline
  Arms: Group C: Normal saline

SUMMARY:
To evaluate the efficacy and safety of intravesical instillation of Lipotoxin for the treatment of IC/BPS

DETAILED DESCRIPTION:
Liposome has been proven able to carry botulinum toxin protein across the cell membrane and effect on urothelial receptors in human overactive bladder. However, the therapeutic duration is limited to 1 month. Intravesical BOTOX injection in patients with interstitial cystitis (IC) can effectively decrease pain, improve bladder capacity and decrease frequency. However, the need of cystoscopic injection limits its wide application.

A total of 100 eligible women with non-ulcer IC will be enrolled to receive intravesical instillation of Lipotoxin containing 80mg liposomes and 200U BOTOX (treatment group), 200U BOTOX in normal saline (N/S) (active control group) or normal saline (placebo control group) single treatment. At least 90 evaluable patients will be included for the final analysis.

All patients should have IC symptoms for at least 6 months, and proven to have grade 2 diffused glomerulations after cystoscopic hydrodistention (HD) within recent 1 year without Hunner's lesion. Patients should not have UTI in recent 12 months, no urinary tract stone. Patients should have been proven free of detrusor overactivity or bladder outlet obstruction. Patients should not receive intravesical hyaluronic acid treatment in recent 6 months, or intravesical Botox injection in recent 12 months. Intravesical instillation of Lipotoxin at OPD and the patient should hold the solution for 2 hours to allow bladder distention. Retreatment with Lipotoxin at 3 months if patient reports ineffective.

Primary end-point is the change of the O'Leary-Sant symptom score (including ICSI and ICPI) from baseline to 1 month after treatment. Secondary endpoints include VAS, daily frequency, nocturia and FBC as record in 3-day voiding diary, Qmax, voided volume, PVR and global response assessment (GRA). Four visits are required at baseline screening (before first treatment), treatment (V1), 2 weeks (V2), 4 weeks (V3, primary end-point) and 12 weeks (V4).

ELIGIBILITY:
Inclusion Criteria:

1. Adults with age of 20 years old or above
2. Patients with symptoms of frequency, urgency, nocturia, and/or bladder pain.
3. Proven to have glomerulations (at least grade 2) by cystoscopic hydrodistention under anesthesia in recent 1 year
4. Free of active urinary tract infection
5. Free of bladder outlet obstruction on enrollment
6. Free of overt neurogenic bladder dysfunction and limitation of ambulation
7. Patient or his/her legally acceptable representative has signed the written informed consent form

Exclusion Criteria:

1. Hunner's lesion proven by cystoscopy
2. Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
3. Patients with bladder outlet obstruction on enrollment
4. Patients with postvoid residual >250ml
5. Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
6. Patients have laboratory abnormalities at screening including: ALT> 3 x upper limit of normal range, AST> 3 x upper limit of normal range; Patients have abnormal serum creatinine level > 2 x upper limit of normal range
7. Patients with any contraindication to be urethral catheterization during treatment
8. Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
9. Myasthenia gravis, Eaton Lambert syndrome.
10. Patients with any other serious disease considered by the investigator not in the condition to enter the trial
11. Patient had received intravesical treatment for IC within recent 1 month
12. Patients participated investigational drug trial within 1 month before entering this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change of the O'Leary-Sant symptom score | Baseline and 1 month
  Change of the O'Leary-Sant symptom score from baseline to 1 month after the treatment day

SECONDARY OUTCOMES:
Net changes of the Visual Analog Scale (VAS) | Baseline and 1 month
  Net changes of the Visual Analog Scale from baseline to 1 month after the treatment day
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net changes of the functional bladder capacity (FBC) | Baseline and 1 month
  Net changes of the functional bladder capacity from baseline to 1 month after the treatment day
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net changes of the voiding frequency at daytime as recorded in 3-day voiding diary | Baseline and 1 month
  Net changes of the voiding frequency at daytime from baseline to 1 month after the treatment day
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net changes of the voiding frequency at night time as recorded in 3-day voiding diary | Baseline and 1 month
  Net changes of the voiding night time from baseline to 1 month after the treatment day
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net Change of the Global response assessment (GRA) | Baseline and 1 month
  Global response assessment (GRA) of therapeutic result by the patient (categorized from -3 to +3, indicating markedly worse to markedly improved) at 3 months after the treatment day.
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net Change of the maximum flow rate | Baseline and 1 month
  Net changes of the maximum flow rate from baseline to 1 month after the treatment day.
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net Change of the voided volume | Baseline and 1 month
  Net changes of the voided volume from baseline to 1 month after the treatment day.
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net Change of the PVR | Baseline and 1 month
  Net changes of the PVR from baseline to 1 month after the treatment day.
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net Change of the urinary nerve growth factor | Baseline and 1 month
  Changes of urinary nerve growth factor from baseline to 1 month after treatment day.
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).
Net Change of the cytokines level | Baseline and 1 month
  Changes of cytokines level from baseline to 1 month after treatment day.
  Safety
  (1) Local adverse event incidences (hematuria, miction pain, UTI, urinary retention).

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddihisst Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD cannot be released unless researchers obtain the approval from the Ethics Committee of the Buddhist Tzu Chi General Hospital, Hualien, Taiwan

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597